CLINICAL TRIAL: NCT00000963
Title: A Randomized Comparative Trial of Two Doses of 2',3'-Dideoxyinosine (ddI) in Children With Symptomatic HIV Infection Who Are Either Unresponsive to Zidovudine and/or Who Are Intolerant to Zidovudine
Brief Title: A Study of Dideoxyinosine (ddI) in HIV-Infected Children Who Have Not Had Success With Zidovudine or Who Cannot Take Zidovudine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 144; 11119 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Evaluation; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Didanosine

INTERVENTIONS:
Drug: Didanosine

SUMMARY:
To evaluate the effectiveness, safety, and tolerance of two doses of didanosine (ddI) in the treatment of children with symptomatic HIV disease who have had to discontinue zidovudine (AZT) because of intolerance and/or who have experienced progressive disease while on AZT.

The progression of immunodeficiency due to HIV infection can be delayed by using AZT. The benefits of AZT in adults with AIDS and severe AIDS-related complex (ARC) appear to last for approximately 12 to 18 months, at which time most patients have progressive deterioration. Recently published literature has described a reduced sensitivity of HIV isolated from patients after prolonged AZT treatment. Although the clinical significance of this is unclear, it makes the development of new antiretroviral drugs important.

DETAILED DESCRIPTION:
The progression of immunodeficiency due to HIV infection can be delayed by using AZT. The benefits of AZT in adults with AIDS and severe AIDS-related complex (ARC) appear to last for approximately 12 to 18 months, at which time most patients have progressive deterioration. Recently published literature has described a reduced sensitivity of HIV isolated from patients after prolonged AZT treatment. Although the clinical significance of this is unclear, it makes the development of new antiretroviral drugs important.

Children who show AZT intolerance and/or progressive disease after 6 months of AZT therapy receive oral ddI at 1 of 2 doses for a minimum of 48 weeks, with a 48-week extension. Patients are seen for clinical and laboratory evaluations at scheduled times during the study. (Per 5/12/92 amendment, new patients will not be enrolled in the pharmacokinetics studies.) Per 10/31/94 amendment: Patients are eligible to receive blinded study drug for an additional 8-16 weeks after the final on-study visit, but no later than 2/15/95.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prophylaxis treatment for Pneumocystis carinii pneumonia (PCP).
* Immunoglobulin.
* Maintenance therapy with amphotericin B (l mg/kg) up to 5 days/week.

Concurrent Treatment:

Allowed:

* Blood transfusions.

Prior Medication:

Allowed:

* Prophylaxis treatment for Pneumocystis carinii pneumonia (PCP).

Patients enrolled in ACTG 128 and ACTG 138 must meet study end points or meet protocol definitions for being permanently off zidovudine (AZT) before enrolling in this study.

* Patients currently enrolled in ACTG 051 who have not reached the study end points but who meet the entry criteria for ACTG 144 may be co-enrolled in ACTG 144.
* Patient or guardian available to give written informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded.

* Hypersensitivity to didanosine (ddI).
* Symptomatic cardiomyopathy.
* Seizures that are not well controlled by ongoing anticonvulsant therapy.
* Symptomatic pancreatitis.
* Grade 1 or higher peripheral neuropathy.
* Active malignancy requiring chemotherapy.

Concurrent Medication:

Excluded:

* Zidovudine (AZT), other antiretroviral agents, biological modifiers, and investigational medications.

Avoid:

* Drugs with potential to cause peripheral neuropathy or pancreatitis.

Patients with the following are excluded:

* Active malignancy requiring concomitant chemotherapy.

Prior Medication:

Excluded:

* Antiretroviral agents other than zidovudine (AZT) or dideoxycytidine (ddC) within 4 weeks of study entry.
* Immunomodulating agents such as interferons, isoprinosine, or interleukin-2 within 2 weeks of entry.
* Any other experimental therapy within 1 week of entry.
* Drugs that have or will cause prolonged neutropenia, significant pancreatitis, significant nephrotoxicity, or peripheral neuropathy within 1 week of entry.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300
Dates: Study Completion 1995-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frenkel LM, Study Chair; Bryson Y, Study Chair; Stiehm R, Study Chair
Locations (52):
- United States (49):
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - Usc La Nichd Crs, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Harbor - UCLA Med. Ctr. - Dept. of Peds., Div. of Infectious Diseases, Torrance, California
  - Univ. of Connecticut Health Ctr., Dept. of Ped., Farmington, Connecticut
  - Yale Univ. School of Medicine - Dept. of Peds., Div. of Infectious Disease, New Haven, Connecticut
  - Children's National Med. Ctr., ACTU, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Emory Univ. School of Medicine, Dept. of Peds., Div. of Infectious Diseases, Atlanta, Georgia
  - Cook County Hosp., Chicago, Illinois
  - Univ. of Illinois College of Medicine at Chicago, Dept. of Peds., Chicago, Illinois
  - Chicago Children's CRS, Chicago, Illinois
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Univ. of Maryland Med. Ctr., Div. of Ped. Immunology & Rheumatology, Baltimore, Maryland
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - UMDNJ - Robert Wood Johnson, New Brunswick, New Jersey
  - St. Joseph's Hosp. & Med. Ctr. of New Jersey, Paterson, New Jersey
  - Children's Hospital at Albany Medical Center, Dept. of Peds., Albany, New York
  - SUNY Downstate Med. Ctr., Children's Hosp. at Downstate NICHD CRS, Brooklyn, New York
  - North Shore-Long Island Jewish Health System, Dept. of Peds., Great Neck, New York
  - Schneider Children's Hosp., Div. of Infectious Diseases, New Hyde Park, New York
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Metropolitan Hosp. NICHD CRS, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Incarnation Children's Ctr., New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - Case CRS, Cleveland, Ohio
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - St. Christopher's Hosp. for Children, Philadelphia, Pennsylvania
  - Med. Univ. of South Carolina, Div. of Ped. Infectious Diseases, Charleston, South Carolina
  - Children's Med. Ctr. Dallas, Dallas, Texas
  - Texas Children's Hosp. CRS, Houston, Texas
  - UW School of Medicine - CHRMC, Seattle, Washington
- Puerto Rico (3):
  - Univ. Hosp. Ramón Ruiz Arnau, Dept. of Peds., Bayamón
  - San Juan City Hosp. PR NICHD CRS, San Juan
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan

REFERENCES:
- [Background] Carey VJ, Yong F, Frenkel L, McKinney R. Enhancing the prognostic value of bodily growth histories in HIV-positive pediatric cohorts. Int Conf AIDS. 1996 Jul 7-12;11(2):134 (abstract no WeC3444)
- [Background] Perrier M, Schwarz T, Gonzalez O, Brounts S. Squamous cell carcinoma invading the right temporomandibular joint in a Belgian mare. Can Vet J. 2010 Aug;51(8):885-7. PMID 21037891